CLINICAL TRIAL: NCT02272166
Title: Effects of Propofol on Early Recovery of Hunger After Ambulatory Surgery Compared With Sevoflurane
Brief Title: Effects of Propofol on Early Recovery of Hunger After Surgery
Acronym: Propo-Faim
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014/088/HP
Record Dates: First submitted 2014-10-15; First posted 2014-10-22 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Ambulatory Surgery; Anesthesia; Energy Expenditure; Food Intake
MeSH Terms: interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- propofol (Active Comparator): Hypnotic used in this arm is exclusively intra-venous propofol.
  Interventions: Drug: propofol
- sevoflurane (Active Comparator): Hypnotic used in this arm is exclusively inhaled sevoflurane.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: propofol
  Other Names: diprivan, 2,6-bis(propan-2-yl)phénol
  Arms: propofol
Drug: Sevoflurane
  Other Names: Sevorane, 1,1,1,3,3,3-hexafluoro-2-(fluorométhoxy)propane
  Arms: sevoflurane

SUMMARY:
Recovery of hunger is a source of comfort for patients after general anesthesia. Moreover, this aspect of post-operative period is often required for discharging patients from hospital after ambulatory surgery. Indeed, this item is part of a multi-parameter score (Chung score) whose validation evaluates patient's ability to return home.

The impact of anesthetics on hunger is largely unknown but few studies suggest an orexigenic effect of propofol compared to halogenated gases. These studies had neither the power nor the methodology to answer the question. The aim of our study is to evaluate the impact of propofol versus sevoflurane on early recovery of hunger after ambulatory surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old women
* American Society of Anesthesiologists (ASA) score 1-2
* Affiliated to a social security system
* Undergoing an ambulatory surgery during more than 15 minutes with general anesthesia and control of upper airways (tracheal intubation or supraglottic mask or facial mask ventilation) for oocytes punction before in vitro fertilization
* General anesthesia occuring between 8 and 10 am with respect of pre-operative fasting rules
* APFEL risk score for nausea and vomiting ≤ 2/4
* Ability to understand and read french
* Signature of understood consent

Exclusion Criteria:

* Other surgery than oocytes punction
* Cognitive dysfunction
* Undernutrition or risk factor of undernutrition (evolutive neoplasia, chronic alcoholism …)
* BMI ≥ 35 kg/m²
* Eating disorders
* Diabetes mellitus
* Chronic treatment with drugs modifying feeding behavior :

  * Benzodiazepines
  * Inhibitors of serotonin reuptake
  * Others
* Non respect of pre-operative fasting rules
* Indication for rapid sequence induction (gastro-oesophageal reflux, absence of gastric emptying …)
* Contraindication to propofol (allergia to propofol, soybean or peanuts, past history of propofol infusion syndrome, unstable cardiovascular disease) or to sevoflurane (past history of malignant hyperthermia, epilepsy or liver disorders after administration of a halogenated anesthetic)
* Pregnant or breastfeeding woman
* Involvement in another clinical trial under 4 previous weeks

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2014-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Time before recovery of hunger after general anesthesia | 1-4 hours
  Time before appearance of of hunger (evaluated by a score above 50/100 mm on analogic visual scale) after the end of hypnotic administration (propofol or sevoflurane).

SECONDARY OUTCOMES:
Feeding comfort | 1-4 hours
  Amount of food intake evaluated by a specific scale
Post operative nausea and vomiting | 1-4 hours
Validation of Chung score | 1-4 hours
  Time needed to obtain a Chung score superior or equal to 9/10, permitting the patient to return home
Change in plasmatic leptin level | 0-3 hours
  Change in plasmatic leptin level (expressed in ng/ml) at the end of anesthesia, one and two hours later, compared with pre-operative value for each patient. Dosage is realized by ELISA method.
Change in plasmatic insulin level | 0-3 hours
  Change in plasmatic insulin level (expressed in microU/ml) at the end of anesthesia, one and two hours later, compared with pre-operative value for each patient. Dosage is realized by ELISA method.
Change in plasmatic ghrelin level | 0-3 hours
  Change in plasmatic ghrelin level (expressed in pg/ml) at the end of anesthesia, one and two hours later, compared with pre-operative value for each patient. Dosage is realized by ELISA method.

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Dureuil, MD-PHD, Study Chair — Departement of Anesthesia, University Hospital, Rouen; Emmanuel BESNIER, MD, Principal Investigator — Departement of Anesthesia, University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

REFERENCES:
- [Derived] Besnier E, Perdrix A, Gillibert A, Selim J, Froemer B, Ghemired A, Berby B, Rives N, Dureuil B, Clavier T, Compere V. Postoperative hunger after outpatient surgery in patients anesthetized with propofol vs sevoflurane: a randomized-controlled trial. Can J Anaesth. 2020 May;67(5):550-559. doi: 10.1007/s12630-020-01584-w. Epub 2020 Jan 29. PMID 31997087